CLINICAL TRIAL: NCT04829422
Title: Multi-center, Prospective, Early Access Program of Lazertinib in Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Patients With T790M Mutation-positive After 1st/2nd Generation EGFR TKIs Therapy to Assess the Safety and Efficacy of Real World Evidence.
Brief Title: Early Access Program of Lazertinib in Republic of Korea
Status: Approved for marketing | Type: Expanded Access
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: LASER-EAP
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — lazertinib

INTERVENTIONS:
Drug: Lazertinib 240 mg — The initial dose of lazertinib 240 mg (3 tablets of 80 mg lazertinib) once daily can be reduced to 160 mg once daily (2 tablets of 80 mg lazertinib) under specific circumstances
  Other Names: Leclaza 240 mg

SUMMARY:
This early access program will be conducted to provide access to Lazertinib for adult patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) with T790M mutation-positive after 1st/2nd generation EGFR TKIs Therapy.

DETAILED DESCRIPTION:
Lazertinib is an oral, highly potent, mutant-selective and irreversible EGFR Tyrosine-kinase inhibitors (TKIs) targets both the T790M mutation and activating EGFR mutations while sparing wild type-EGFR.

This is a Multi-center, Prospective, Early Access Program of Lazertinib in locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) patients with T790M mutation-positive after 1st/2nd generation EGFR TKIs therapy to assess the safety and efficacy of real world evidence as second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 19 years
* Patients who have written consent for use of personal and medical information for the study purpose
* Patients who are prescribed and administered with approved indication for Lazerinib in Korea and not been treated with Lazertinib previously.

Exclusion Criteria:

* Patients with hypersensitivity to Lazertinib or its any ingredients
* Patients who belong to contraindication listed on lazertinib label in Korea
* Patients who are treated for an indication not approved for the use of Lazertinib
* Women who are pregnant or may possibly become pregnant

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult